CLINICAL TRIAL: NCT06003140
Title: Efficacy of Low-cost Warming Mattress Celsi Warmer for the Management of Hypothermic Newborns at the Lagos University Teaching Hospital in Lagos, Nigeria
Brief Title: Efficacy of Celsi Warmer for the Management of Hypothermic Newborns at the Lagos University Teaching Hospital in Lagos, Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Collaborators: University of Lagos, Nigeria (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FY2023-69
Record Dates: First submitted 2023-05-31; First posted 2023-08-21 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Neonatal Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypothermic Neonates (90) (Experimental): A trained study clinician will attach the Celsi Warmer temperature sensor to the abdomen and secure it with the abdominal belt according to the device's instruction manual (such that the temperature sensor is positioned using a vertical line from the mid-clavicular line and just below the ribs). The time of sensor placement will be recorded.
  Interventions: Device: Celsi Warmer

INTERVENTIONS:
Device: Celsi Warmer — A trained study clinician will attach the Celsi Warmer temperature sensor to the abdomen and secure it with the abdominal belt according to the device's instruction manual (such that the temperature sensor is positioned using a vertical line from the mid-clavicular line and just below the ribs). The time of sensor placement will be recorded.

SUMMARY:
The prevalence of hypothermia across low-resource settings is high, especially in countries with high neonatal mortality rates. If left untreated, hypothermia can additionally result in a significant comorbidity, and has been linked to a reduction in the effectiveness of treatment for other newborn conditions. Effective thermal care for hypothermic newborns is not widely available in low-resource settings due to cost of consumables and spare parts. In this study, the research team wish to evaluate the efficacy of a novel neonatal warming mattress in treating hypothermic newborns. Warming mattress, 'Celsi Warmer', has been developed by Rice 360 Institute for Global Health Technologies, in conjunction with African clinicians, to be a robust, low-cost, and easy-to-use warming mattress which can address the challenges of hypothermia. This is a single-arm, non-randomized, prospective intervention study. Up to 90 eligible infants at the neonatal wards of the Lagos University Teaching Hospital will be recruited to evaluate the efficacy of Celsi Warmer in rewarming hypothermic newborns. Infants temperature will be monitored during thermal intervention and the performance of the device will be evaluated. The temperatures of each infant will be compared before, during, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Any neonate who:

1. Is currently being treated at study location,
2. Is an inborn admission to the neonatal ward,
3. Whose parents or guardians provided informed consent,
4. Whose parents or guardians providing informed consent are 18 years old or older,
5. Has a current weight of greater than or equal to 1.0 kg and less than or equal to 4.0 kg,
6. Has been identified as in need of thermal care defined as having a moderate to severe hypothermic temperature (32.0-36.0 °C) as the last temperature recorded in hospital chart, or during recruitment procedures; and
7. is unable to be enrolled in Kangaroo Mother Care (KMC) for reasons including, but not limited to: a. Mother/guardian unable or unavailable to provide KMC b. Under observation in the Neonatal Intensive Care Unit (NICU) before transfer to KMC c. No space in KMC d. Clinician's discretion;
8. May be receiving other medical treatments, including but not limited to, Continuous Positive Airway Pressure (CPAP), oxygen therapy, intravenous (IV) fluids, management and monitoring of common newborn conditions such as hypoglycemia, and/or hyperbilirubinemia.

Exclusion Criteria:

1. Requires mechanical ventilation;
2. Is deemed in need of intensive care by the hospital staff who is providing care, including but not limited to: a. neonates with severe anemia and/or any suspected hematological disorders, and/or b. Neonates with obvious congenital anomalies, and/or c. neonates suspected with hypo/hyperthyroidism or any hormonal disorders;
3. has been diagnosed with birth asphyxia;
4. Presents a condition that precludes the use of the temperature sensor and/or abdominal belt including but not limited to, known umbilical cord infection, known skin infection;
5. Whose clinician presents concerns about their participation;
6. Is receiving treatment that participation in the study would interfere with (e.g. transferring to KMC).

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-21 (Estimated); Study Completion 2024-10-21 (Estimated)

PRIMARY OUTCOMES:
Broad Objective - Comparison to the Gold Standard of Rewarming Hypothermic Newborns | 1 year
  To evaluate the clinical efficacy and safety of the Celsi Warmer in rewarming hypothermic newborns by comparing the Celsi Warmer's accuracy in measuring neonatal temperature compared to the gold standard, axillary temperature readings.

SECONDARY OUTCOMES:
Efficacy of the Device | 1 year
  To assess the performance of the Celsi Warmer in rewarming hypothermic newborns by measuring the incidence of attainment of normothermia (36.5-37.5°C)
Safety of the Device - Rate of Temperature Increase | 1 year
  To measure the infant's rate of temperature (°C) increase through thermoregulatory intervention.
Safety of the Device - Local effect of the Abdominal Belt | 1 year
  To evaluate the local effect of the abdominal belt on newborn's skin by looking at any evidence of skin irritation
Safety of the Device - Incidence of Hyperthermia | 1 year
  To evaluate any incidence of hyperthermia (>37.5°C) during the thermoregulation intervention.
Safety of the Device - Incidence of Rebound Hypothermia | 1 year
  To report any incidence of rebound hypothermia ( < 36.5°C) (post-intervention hypothermia) up to 72 hours from the initial encounter

CONTACTS AND LOCATIONS:
Overall Officials: Chinyere Ezeaka, MBBS, MPH, Principal Investigator — College of Medicine, University of Lagos, Lagos, Nigeria
Locations (1):
- University of Lagos, Lagos, Nigeria, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar V, Shearer JC, Kumar A, Darmstadt GL. Neonatal hypothermia in low resource settings: a review. J Perinatol. 2009 Jun;29(6):401-12. doi: 10.1038/jp.2008.233. Epub 2009 Jan 22. PMID 19158799
- [Background] Carns J, Kawaza K, Quinn MK, Miao Y, Guerra R, Molyneux E, Oden M, Richards-Kortum R. Impact of hypothermia on implementation of CPAP for neonatal respiratory distress syndrome in a low-resource setting. PLoS One. 2018 Mar 15;13(3):e0194144. doi: 10.1371/journal.pone.0194144. eCollection 2018. PMID 29543861
- [Background] Mullany LC. Neonatal hypothermia in low-resource settings. Semin Perinatol. 2010 Dec;34(6):426-33. doi: 10.1053/j.semperi.2010.09.007. PMID 21094417
- [Background] Lunze K, Bloom DE, Jamison DT, Hamer DH. The global burden of neonatal hypothermia: systematic review of a major challenge for newborn survival. BMC Med. 2013 Jan 31;11:24. doi: 10.1186/1741-7015-11-24. PMID 23369256
- [Background] Cavallin F, Calgaro S, Brugnolaro V, Seni AHA, Muhelo AR, Da Dalt L, Putoto G, Trevisanuto D. Impact of temperature change from admission to day one on neonatal mortality in a low-resource setting. BMC Pregnancy Childbirth. 2020 Oct 23;20(1):646. doi: 10.1186/s12884-020-03343-7. PMID 33097025
- [Background] Ogunlesi TA, Ogunfowora OB, Ogundeyi MM. Prevalence and risk factors for hypothermia on admission in Nigerian babies <72 h of age. J Perinat Med. 2009;37(2):180-4. doi: 10.1515/JPM.2009.014. PMID 18684103